CLINICAL TRIAL: NCT07053488
Title: A Phase 1/2, Open-Label, Single-Arm Study to Evaluate the Safety, Immunogenicity Reduction, Transplant Function, and Feasibility of Ex Vivo CRISPR-Cas9 Gene-Edited Donor Liver Transplantation Targeting HLA Class I (HLA-A, HLA-B) and Class II (Via CIITA) Genes.
Brief Title: CRISPR-Edited HLA Donor Liver Transplant to Reduce Rejection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AMERICAN ORGAN TRANSPLANT AND CANCER RESEARCH INSTITUTE LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOTCRI-102
Record Dates: First submitted 2025-06-08; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Liver Diseases; Liver Cancer; Liver Cirrhosis; Liver Failure; Liver Metastases; Liver Transplant Rejection; Liver Steatoses
Keywords: End-Stage Liver Disease requiring transplantation; Prevention of Allograft Rejection in Liver Transplantation; CRISPR-Cas9; Gene Editing; Liver Transplant; Organ Transplantation; Immunogenicity Reduction; HLA Knockout; Hypoimmunogenic Graft; Allograft Rejection; Universal Donor Organ
MeSH Terms: conditions — Liver Diseases; Liver Neoplasms; Liver Cirrhosis; Liver Failure; Fatty Liver

STUDY DESIGN:
Intervention Model Description: All enrolled participants receive the experimental intervention (no control arm). The trial is Open-Label (no blinding) and designed as a combined Phase 1/2 study focusing on safety and preliminary efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRISPR-Edited Donor Liver Transplant (Experimental): Participants undergo orthotopic liver transplantation using a donor liver that has been ex vivo gene-edited by CRISPR-Cas9 to knock out HLA class I (A, B) and class II (via CIITA) genes. There is no comparator arm; outcomes will be compared to historical norms of unedited transplants for context.
  Interventions: Biological: Ex Vivo CRISPR-Cas9 Gene Editing of Donor Liver

INTERVENTIONS:
Biological: Ex Vivo CRISPR-Cas9 Gene Editing of Donor Liver — Donor liver tissue is perfused outside the body with a CRISPR-Cas9 RNP complex targeting HLA-A, HLA-B, and CIITA, to create a hypoimmunogenic graft. After confirming successful gene knockout, the liver is transplanted into the patient following standard surgical techniques. Post-operative care includes routine immunosuppressive therapy with planned adjustments based on the patient's tolerance and evidence of graft immunogenicity.

SUMMARY:
This early-phase clinical trial will assess the use of ex vivo CRISPR-Cas9 genome editing on donor liver grafts to reduce immunogenicity before transplantation. Donor livers will have HLA-A and HLA-B genes knocked out, and HLA class II expression disabled (by targeting the CIITA transactivator gene), aiming to create a "hypoimmunogenic" organ less prone to rejection. The edited liver is then transplanted into patients with end-stage liver disease. The primary focus is on safety and feasibility - determining whether a CRISPR-edited liver can be transplanted successfully and function normally - as well as evaluating reductions in immune response (acute rejection, anti-donor T cell activation) and graft function over time.

DETAILED DESCRIPTION:
Organ transplant rejection is primarily driven by immune recognition of donor HLA (human leukocyte antigen) molecules as foreign. Mismatches in HLA-A and HLA-B (class I) in particular are strongly immunogenic and can provoke T-cell mediated graft rejection. HLA class II molecules (HLA-DR, DQ, DP), expressed on donor antigen-presenting cells, can also activate CD4⁺ T cells and contribute to rejection. Current therapy relies on immunosuppressive drugs, which carry significant risks. Preclinical research has shown that genetically "erasing" HLA molecules from donor cells can blunt immune responses: for example, cells with HLA-A, HLA-B, and HLA-DR knocked out via CRISPR elicited little to no T cell proliferation in vitro, indicating greatly reduced immunogenicity. Similarly, in xenotransplant models, triple knockout of genes (including class I and the class II regulator CIITA) in donor animals significantly weakened human T-cell activation and prolonged graft survival. These findings provide a strong rationale that an HLA-edited donor organ could evade the human immune system to a large extent, potentially reducing or delaying rejection.

Gene-Editing of Donor Liver Ex Vivo: In this trial, deceased-donor livers will undergo ex vivo CRISPR-Cas9 genome editing prior to transplantation. The editing targets are HLA-A and HLA-B (to eliminate the major class I alloantigens) and CIITA (class II transactivator, whose knockout abolishes HLA-DR/DQ/DP expression on donor cells). By knocking out HLA-A and -B, while leaving HLA-C expression intact, the goal is to remove the most immunogenic class I molecules yet maintain some HLA presence to mitigate natural killer cell "missing-self" responses. Disabling CIITA will prevent expression of HLA class II proteins, thus reducing CD4⁺ T cell activation against the graft. The CRISPR editing is performed during machine perfusion of the donor liver (a period in which the organ is kept alive outside the body). A CRISPR-Cas9 ribonucleoprotein (Cas9 enzyme complexed with guide RNAs for HLA-A, HLA-B, and CIITA) is delivered into the liver tissue through the perfusion circuit. Editing takes place ex vivo, avoiding direct in vivo gene therapy to the recipient. Before transplantation, the graft is assessed for successful gene knockout (for example, by biopsy immunostaining or flow cytometry to confirm absence of HLA-A/B/DR on the cell surface). Only livers with confirmed high-efficiency editing (e.g. >90% target gene disruption) are used for transplant to ensure maximal immune-evasion benefit.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 16-85 (inclusive) with end-stage liver disease or acute liver failure who are eligible for liver transplantation.
* Require a liver transplant and have been allocated a donor liver graft (from a deceased donor) that will be used in the study after gene editing.
* No immediately available fully HLA-matched donor (since the study targets patients who would otherwise receive an HLA-mismatched organ; standard allocation generally does not consider HLA matching for liver, so most patients will qualify).
* Medically suitable for transplant surgery and able to tolerate standard immunosuppressive therapy (no contraindications to transplant such as uncontrolled infection or other active serious disease that would preclude surgery).
* Informed Consent: Able to understand the investigational nature of the trial and provide written informed consent. Patients (and their legal representatives if applicable) must consent to the use of a genetically modified organ and to long-term follow-up including multiple biopsies and immune monitoring.
* Willingness to comply with all study procedures and availability for the duration of follow-up (including frequent monitoring visits).

Exclusion Criteria:

* Active uncontrolled infection (e.g., sepsis, active tuberculosis) that would severely increase transplant risk or confound interpretation of immune-related outcomes.
* Uncontrolled HIV or chronic viral infections that are not well-managed. (Note: Patients with hepatitis B or C may be included if adequately treated or under control, as these are common in liver failure, but such patients should not have active, replicating virus at transplant if possible.)
* Multi-organ transplant requirement: Patients needing more than a liver alone (e.g., liver-kidney dual transplant) are excluded, as the trial is only evaluating single organ (liver) outcomes.
* Pregnancy or breastfeeding: Female participants of childbearing potential must have a negative pregnancy test prior to transplant and must agree to use effective contraception. The effects of a gene-edited organ transplant on a fetus/infant are unknown, and immunosuppressive drugs can also harm a pregnancy.
* Severe concurrent illness not related to liver disease that would limit survival to <1 year or make the patient an unsuitable candidate (e.g., advanced heart failure, uncontrolled diabetes with complications, etc.).
* Allergy or hypersensitivity to study-related products: If any components used in the ex vivo gene editing (such as a specific vehicle or enzyme) have known severe allergies in the recipient, they will be excluded. (For instance, although unlikely, if a patient had a documented severe immune reaction to Streptococcus pyogenes Cas9 or similar proteins, they would not be enrolled.)
* Inability to follow the protocol or comply with follow-up: this includes psychiatric, social or logistical factors that would prevent adhering to the intense monitoring schedule (for example, lack of reliable transportation or support).

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-18 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade ≥3 Treatment-Emergent Adverse Events (TEAEs) | Day 1 to Day 90
  Number of participants experiencing ≥1 CTCAE v5.0 Grade 3-5 TEAE judged related to the gene-edited liver transplant procedure
Feasibility of Ex Vivo HLA Gene Editing | Day1 to Day 90
  Proportion of donor livers that achieve the desired editing criteria (e.g., >90% knockout efficiency of HLA-A/B and abolition of class II expression) and are successfully transplanted into recipients. Feasibility is further indicated by the absence of technical issues during organ editing and transplantation.
Graft Failure Rate at Day 90 | Day1 to Day 90
  Proportion of participants requiring re-transplant, graft explant, or returning to listing due to primary non-function.Unit of Measure :Participants with graft failure (n, %)

SECONDARY OUTCOMES:
Incidence of Acute Rejection at 6 and 12 Months | Day 1 - Month 12
  The proportion of patients experiencing biopsy-confirmed acute cellular rejection episodes within 6 months and within 12 months post-transplant. The severity of rejection (graded by standard criteria) and response to treatment will also be recorded. A lower-than-expected rejection rate or milder rejection would indicate a successful immunogenicity reduction.
Immunologic Markers of Alloreactivity | Day 1 - Month 12
  Levels of anti-donor HLA antibodies in recipient blood (donor-specific antibodies, DSA) and T-cell alloimmune reactivity (e.g., in vitro mixed lymphocyte reaction or ELISPOT assays against donor cells) at 3, 6, and 12 months. We will compare these immunologic markers to baseline and to typical post-transplant profiles. We hypothesize that patients with edited grafts will show attenuated T cell responses to donor antigens.
Graft Survival and Function at 1 Year | Day 1 - Month 12
  Number of patients with the original transplanted liver surviving at 12 months with no graft loss.
Patient Survival at 1 Year | 12 months
  Overall survival of participants at 1 year post-transplant.
Immunosuppression Reduction Feasibility | 12 months
  Among patients with stable graft function, ability to taper down immunosuppressive therapy by 6-12 months post-transplant without precipitating rejection. This will be measured by the proportion of patients successfully maintaining graft health on reduced immunosuppressant dosage or simpler regimen.
Off-target Effects Assessment | 24 months
  trial will evaluate any evidence of off-target gene editing effects manifesting in the graft (for example, unexpected histological changes, or aberrant liver function that could hint at unintended gene disruptions). Genomic analyses of edited tissue will be done to characterize off-target mutation frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Health Science Center (PKUHSC), Beijing, Changping, China

IPD SHARING:
Plan to Share IPD: No